CLINICAL TRIAL: NCT05399680
Title: Evaluation of Safety and Efficacy of the S.M.A.R.T. RADIANZ™ Vascular Stent System in the Treatment of Iliac and Femoropopliteal Lesions Via Transradial Access
Acronym: RADIANCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Collaborators: Qserve (Industry); NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P21-7701
Record Dates: First submitted 2022-02-22; First posted 2022-06-01 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Interventional (Experimental): Treatment with SMART RADIANZ, BRITE TIP RADIANZ and SABERX RADIANZ devices
  Interventions: Device: S.M.A.R.T. RADIANZ™ Vascular Stent System; Device: BRITE TIP RADIANZ™ Guiding Sheath; Device: SABERX RADIANZ™ PTA Balloon Catheter

INTERVENTIONS:
Device: S.M.A.R.T. RADIANZ™ Vascular Stent System — The S.M.A.R.T. RADIANZ™ Vascular Stent System is designed to deliver the S.M.A.R.T.™ self-expanding stent (S.M.A.R.T.™ stent) to the iliac arteries, superficial femoral arteries and/or proximal popliteal arteries using a 6F (2.0 mm) sheathed delivery system introduced through the radial artery.
Device: BRITE TIP RADIANZ™ Guiding Sheath — BRITE TIP RADIANZ™ is a catheter guiding sheath that facilitates percutaneous entry of an intravascular device into the peripheral vasculature through the radial artery.
Device: SABERX RADIANZ™ PTA Balloon Catheter — SABERX RADIANZ™ is a catheter with a distal inflatable balloon.

SUMMARY:
The primary objective of this clinical investigation was to evaluate acute safety and efficacy of the S.M.A.R.T. RADIANZ™ Vascular Stent System, when used with the BRITE TIP RADIANZ™ Guiding Sheath and SABERX RADIANZ™ PTA Balloon Catheter, to deploy the S.M.A.R.T.™ Nitinol Stent, in the treatment of patients with obstructive iliac or femoropopliteal arterial disease via radial artery access.

DETAILED DESCRIPTION:
RADIANCY was an acute, multi-center, single-arm, non-randomized, prospective, pivotal (pre-market) clinical study, whose primary objective was to evaluate acute safety and efficacy of the S.M.A.R.T. RADIANZ™ Vascular Stent System, when used with the BRITE TIP RADIANZ™ Guiding Sheath and SABERX RADIANZ™ PTA Balloon Catheter, to deploy the S.M.A.R.T.™ self-expanding stent in the treatment of patients with obstructive iliac or femoropopliteal arterial disease via transradial artery access. The study enrolled 151 subjects, 22 of which were enrolled as "roll-in" subjects, at 12 investigational sites across Europe. These subjects were followed up to 30 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following inclusion criteria to be enrolled in the study:

ALL patients must meet the following criteria prior to enrollment:

1. Age ≥ 18 years
2. For women of child-bearing potential, a negative pregnancy test within seven (7) days prior to the index procedure
3. Symptomatic leg ischemia or ischemic ulcerations that do NOT exceed digits of the foot (Rutherford/Becker Classification category 2, 3, 4 or 5)
4. Palpable radial artery with diameter ≥ 2.5 mm, as assessed by duplex ultrasound
5. Eligibility for standard surgical repair, if necessary
6. A patient who requires a coronary intervention should have it performed at least seven (7) days prior to treatment of the target lesion
7. The patient must provide documented informed consent and any other documented authorization, as required, prior to initiation of the study procedure
8. Per Investigator assessment, the patient is willing and able to be followed up to 30 days post-procedure for evaluation and complete all required assessments per the study protocol.

   Inclusion criteria 9 and 10 AND 11a through 14a OR 11b through 16b (whichever is applicable) would be assessed via baseline angiography performed at the time of index procedure:
9. The Investigator has assessed that the patient is a suitable candidate (i.e, meets all inclusion criteria and none of the exclusion criteria), for treatment of a lesion in the iliac, superficial femoral and/or proximal popliteal arteries via transradial approach and is eligible for conversion from a transradial to transfemoral approach, if it becomes necessary.
10. The guidewire is across the target lesion(s) and located intraluminally within the distal vessel following a transradial approach

Patients whose target lesion is in the iliac artery must meet these additional criteria prior to enrollment:

11a. A single de novo or restenotic lesion ≥ 50% stenosis in the common and/or external iliac artery

12a. Stenotic lesion (one long or multiple serial/tandem lesions) less than or equal to 100 mm, by visual assessment, within or across the common or external iliac arteries. The stenosis must be treatable with no more than two stents (while minimizing stent overlap)

13a. Reference vessel diameter (RVD) ranging from 4.0 to 9.0 mm by visual assessment

14a. Angiographic evidence of a patent profunda or superficial femoral artery in the diseased (target) limb

Patients whose target lesion is in the SFA and/or PPA must meet these additional criteria prior to enrollment:

11b. A single de novo or restenotic lesion ≥ 50% stenosis in the SFA and/or PPA

12b. Stenotic lesion (one long or multiple serial/tandem lesions) less than or equal to 150 mm, by visual assessment, within or across the SFA and/or PPA. The stenosis must be treatable with no more than two stents (while minimizing stent overlap)

13b. RVD ranging from 4.0 to 7.0 mm by visual assessment

14b. All lesions are to be located at least three centimeters proximal to the superior edge of the patella

15b. Patent infrapopliteal artery, i.e., single vessel runoff or better with patency (<50% stenosis) of at least one of three vessels to the ankle or foot

16b. Adequate aortoiliac or common femoral "inflow" (defined as < 30% stenosis after PTA or stenting) prior to treatment of the target lesion (defined as < 30% stenosis after PTA or stenting) prior to treatment of the target lesion

Exclusion Criteria:

Patients will be excluded if ANY of the following exclusion criteria apply:

1. The patient has had/experienced any prior intervention/treatment to the target vessel within 90 days prior to enrollment (e.g., previously implanted graft in the aorta or target vessel; stroke; cryoplasty, laser or atherectomy; abdominal aortic aneurysm or aneurysm of the iliac, superficial femoral or popliteal artery).
2. Previously deployed stent at the site of the target lesion
3. The patient has post-surgical stenosis and anastomotic suture treatments of the target vessel
4. Requires general anesthesia for percutaneous transluminal angioplasty (PTA) and/or the stenting procedure
5. Use of mechanical devices on or thrombolysis of the target vessel within 72 hours prior to the index procedure without complete resolution of the thrombus
6. The patient is receiving any form of dialysis.
7. The patient is receiving any form of immunosuppressant therapy.
8. Planned amputation
9. Established vasospastic disease
10. Glomerular filtration rate (GFR) < 30 mL/min within 7 days prior to the index procedure
11. The patient has a history of neutropenia, coagulopathy, and/or thrombocytopenia.
12. Thrombophlebitis, uremia, or deep venous thrombus, within past 30 days prior to the index procedure
13. Bleeding diathesis
14. Known allergies or intolerance to antiplatelet, anticoagulant or thrombolytic medications including but not limited to aspirin, clopidogrel bisulfate (Plavix®), ticlopidine (Ticlid®) or heparin that cannot be medically managed.
15. Known allergy or intolerance to Nitinol (nickel titanium)
16. Known allergy to contrast agent that cannot be medically managed before treatment with steroids and/or antihistamines.
17. Known or suspected active infection at the time of the index procedure.
18. Patient is currently participating in another investigational drug or medical device study that has not completed primary endpoint(s) evaluation or clinically interferes with the endpoints from this study or is planning to participate in such a study prior to their completion of this study.
19. Patient has had a major surgical or interventional procedure unrelated to this study within 30 days prior to enrollment or is anticipated/planned to have such a procedure within 30 days after enrollment.

    Exclusion criteria 20 through 25 would be assessed via baseline angiography performed at the time of index procedure:
20. Significant vessel tortuosity or other parameters prohibiting access to the lesion or 90° tortuosity which would prevent delivery of the stent device
21. Noted perforation of the target vessel
22. Stent placement required across or within 0.5 cm of the SFA/profunda femoris artery (PFA) bifurcation
23. Cases of chronic total occlusion/in-stent restenosis/severe calcification in which there is pre-determined inability to treat the target lesion with a single stent, or procedures pre-determined to require stent-in-stent placement to obtain patency
24. Presence of thrombus prior to crossing the lesion
25. Successful PTA treatment of a target lesion in the SFA/PPA (defined as < 50% stenosis after PTA treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Austria (4):
  - Univ Klinikum LKG Graz, Graz
  - Klinikum Klagenfurt am Wörtherse, Klagenfurt
  - Hanusch Krankenhaus, Vienna
  - Univ.-Klinik für Innere Medizin II, Vienna
- A.Z. Sint-Blasius Hospital-Dendermonde, Dendermonde, Belgium
- France (4):
  - Hospital Ambroise Pare, Boulogne-Billancourt
  - Groupe Hôpital Paris St Joseph, Paris
  - Clinique Rhena, Strasbourg
  - Clinique Pasteur, Toulouse
- Maria Cecilia Hospital, Cotignola, Italy
- Hosp Univ. de Guadalajara, Guadalajara, Spain
- Kantonsspital Winterthur, Winterthur, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 151 enrolled subjects were enrolled between June 29, 2022 and September 22, 2023 at 12 institutions/hospitals across 6 European countries.
Pre-assignment Details: Of the 151 total enrolled subjects, 129 subjects belonged to the main cohort while the remaining 22 subjects belonged to a roll-in cohort.
  The outcomes presented in this record are for EACH of the two cohorts in the Participant Flow, Baseline Characteristics and Adverse Events modules and for the MAIN cohort alone in all other modules (i.e., Outcome Measures).
Groups:
- Main Cohort: All enrolled subjects were planned to be treated with the SMART RADIANZ, BRITE TIP RADIANZ and SABERX RADIANZ devices.
  The S.M.A.R.T. RADIANZ™ Vascular Stent System is designed to deliver the S.M.A.R.T.™ self-expanding stent (S.M.A.R.T.™ stent) to the iliac arteries, superficial femoral arteries and/or proximal popliteal arteries using a 6F (2.0 mm) sheathed delivery system introduced through the radial artery.
  BRITE TIP RADIANZ™ is a catheter guiding sheath that facilitates percutaneous entry of an intravascular device into the peripheral vasculature through the radial artery.
  SABERX RADIANZ™ is a catheter with a distal inflatable balloon.
- Roll-in Cohort: A subgroup of 22 subjects, consisting of the first two (2) enrolled subjects at each study site (as applicable), constituted the "roll-in" cohort for the study. Such subjects were pre-specified as "roll-in" subjects prior to their enrollment and met all criteria for enrollment, however, they were also followed up and evaluated up to 30 days post-procedure only for safety and not included in any primary endpoint analyses.
Period: Overall Study
Arm/Group | Main Cohort | Roll-in Cohort
Started | 129 | 22
Completed | 128 | 21
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Main Cohort: Treatment with SMART RADIANZ, BRITE TIP RADIANZ and SABERX RADIANZ devices
- Roll-in Cohort: Treatment with SMART RADIANZ, BRITE TIP RADIANZ and SABERX RADIANZ devices
  A subgroup of 22 subjects, consisting of the first two (2) enrolled subjects at each study site (as applicable), constituted the "roll-in" cohort for the study. Such subjects were pre-specified as "roll-in" subjects prior to their enrollment and met all criteria for enrollment, however, they were also followed up and evaluated up to 30 days post-procedure only for safety and not included in any primary endpoint analyses.
- Total: Total of all reporting groups
Arm/Group | Main Cohort | Roll-in Cohort | Total
Number analyzed (Participants) | 129 | 22 | 151
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.23 (9.44) | 68.45 (8.90) | 68.26 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 3 | 37
  Male | 95 | 19 | 114
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 43 | 8 | 51
  Italy | 17 | 2 | 19
  France | 65 | 8 | 73
  Spain | 4 | 2 | 6
  Switzerland | 0 | 1 | 1
  Belgium | 0 | 1 | 1
Medical History [Count of Participants; unit: Participants] — Smoking Unknown represents cases in which the investigator was unable to confirm whether the subjects had a history of smoking.
  Participants
    COPD | 15 | 4 | 19
    Chronic Renal Failure | 4 | 4 | 8
    Diabetes Mellitus | 39 | 5 | 44
    Heart Failure | 6 | 1 | 7
    Hypercholesterolemia | 93 | 16 | 109
    Hypertension | 98 | 19 | 117
    Peripheral Artery Disease | 96 | 15 | 111
    Previous Cerebrovascular Accident | 7 | 1 | 8
    Previous Myocardial Infarction | 9 | 1 | 10
    Smoking | 91 | 18 | 109
    Smoking Unknown | 3 | 1 | 4
Physical Examination Condition [Count of Participants; unit: Participants]
  Peripheral Artery Disease Symptoms | 129 | 21 | 150
  Claudication Symptoms | 127 | 20 | 147
  Muscle Plain with Exercise | 110 | 17 | 127
  Critical Limb Symptoms | 12 | 3 | 15
  Pain at Rest | 13 | 1 | 14
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 170.48 (8.30) | 172.5 (9.02) | 170.77 (8.41)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 77.01 (14.33) | 82.78 (15.42) | 77.85 (14.59)
Rutherford Class [Count of Participants; unit: Participants] — Rutherford Classification scores range from 0 to 6 with lower scores indicative of better outcomes. Participants were staged/graded clinically by Investigator assessment.
  Participants
    Class 2 - moderate claudication | 46 | 5 | 51
    Class 3 - Severe Claudication | 71 | 16 | 87
    Class 4 - Ischemic Rest Pain | 6 | 0 | 6
    Class 5 - Minor tissue loss-non healing ulcer, focal gangrene with diffuse pedal ischemia | 6 | 1 | 7
Pre-Procedure Stenosis Percent [Mean (Standard Deviation); unit: Percent] — Pre-Procedure Stenosis Percent is the percentage of stenosis in the target vessel that is assessed from the angiogram taken during the index procedure and prior to treatment with any of the study devices.
  Percent
    Reported by Sites | 82.50 (11.06) | 81.27 (12.81) | 81.28 (11.58)
    Reported by Core Lab | 57.56 (25.46) | 58.05 (29.21) | 57.63 (25.94)
Target Lesion Location - Core Lab Reported [Count of Participants; unit: Participants]
  Common iliac artery | 52 | 8 | 60
  Common iliac artery, External iliac artery | 8 | 6 | 14
  Common iliac artery, Superficial femoral artery | 0 | 0 | 0
  External iliac artery | 32 | 3 | 35
  External iliac artery, Superficial femoral artery | 0 | 0 | 0
  Proximal popliteal artery | 0 | 1 | 1
  Superficial femoral artery | 36 | 3 | 39
  Not Stated | 1 | 1 | 2
Lesion Length Characteristic - Core Lab Reported [Mean (Standard Deviation); unit: mm] | 47.58 (44.32) | 54.32 (47.68) | 48.72 (44.78)
Calcification Category - Core Lab Reported [Count of Participants; unit: Participants]
  Severe | 50 | 14 | 64
  Non-Severe | 26 | 2 | 28
  No calcification | 48 | 6 | 54
  Not Stated | 5 | 0 | 5
Radial Artery Diameter by Ultrasound - Site Reported (mm) [Mean (Standard Deviation); unit: mm] — Population: Missing data
  mm
    number analyzed (Participants) | 127 | 22 | 149
    (all) | 3.10 (0.65) | 2.94 (0.45) | 3.07 (0.63)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence Rate of Radial Access Site Complications (Primary Safety Outcome)
Description: Occurrence rate of CEC-adjudicated, major radial access site complications attributed to study device or procedure through time of hospital discharge.
Time Frame: From the time of sheath introduction through the radial artery (start time of procedure) through time of discharge (within ~48 hours of end time of procedure) or study exit, whichever comes first
Population: Intent-to-treat population of the main cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 129
Participants | 0

2. Primary Outcome: Technical Success of Using the S.M.A.R.T. RADIANZ™ Vascular Stent System (Primary Efficacy Outcome)
Description: Technical success at the conclusion of the index procedure, defined as successful insertion of the S.M.A.R.T. RADIANZ™ Vascular Stent System into the peripheral vasculature through the radial artery, successful deployment of the study device (S.M.A.R.T.™ stent) at the intended location, and successful withdrawal of the delivery system without conversion from radial to femoral artery access.
Time Frame: From the time of insertion to the time of withdrawal of the SMART RADIANZ Vascular Stent System through the radial access artery, within the same day or 24 hours from the procedure start time
Population: Intent-to-treat population of the main cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 123
Participants | 122

3. Secondary Outcome: Device Deficiencies Through 30 Days Post-Procedure
Description: For each of the three (3) devices, peri-procedural (within 30 days post-index procedure) rate of device deficiencies
Time Frame: From the time of first use/handling of the device to 30 days from date of index procedure or study exit, whichever comes first
Population: Intent to Treat population of the main cohort. Use of the SMART RADIANZ and SABERX RADIANZ devices was not attempted in all 129 main cohort subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 129
Participants
  BRITE TIP RADIANZ | 1
  SMART RADIANZ: number analyzed (Participants) | 123
  SMART RADIANZ | 1
  SABERX RADIANZ: number analyzed (Participants) | 128
  SABERX RADIANZ | 0

4. Secondary Outcome: Adverse Events Through 30 Days Post-Procedure
Description: Peri-procedural (within 30 days post-index procedure) rate of adverse events
Time Frame: From the time of introduction of the sheath through the radial access artery to 30 days from date of index procedure or study exit, whichever comes first
Population: Intent to Treat population of the main cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 129
Participants | 24

5. Secondary Outcome: Death, Index Limb Amputation and TLR Through 30 Days Post-Procedure
Description: Peri-procedural (within 30 days post-index procedure) rate of death, index limb amputation and target lesion revascularization
Time Frame: as for outcome 4
Population: Intent to Treat population of the main cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 129
Participants
  Death | 0
  Index Limb Amputation | 1
  Target Lesion Revascularization | 0

6. Secondary Outcome: Procedural Complications Through 30 Days Post-Procedure
Description: Peri-procedural (within 30 days post-index procedure) rate of procedural complications
Time Frame: as for outcome 4
Population: Intent to Treat population of the main cohort. The number analyzed is less than 129 in some of the rows below due to the fact that SMART RADIANZ and SABERX RADIANZ devices were not attempted to be used in all 129 main cohort subjects and due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 129
Participants
  No Conversion from Radial Artery | 128
  BRITE TIP RADIANZ Insertion | 129
  Guidewire Across Target Lesion | 129
  SABERX RADIANZ Insertion | 128
  Balloon Inflation: number analyzed (Participants) | 113
  Balloon Inflation | 113
  S.M.A.R.T. RADIANZ Insertion: number analyzed (Participants) | 123
  S.M.A.R.T. RADIANZ Insertion | 123
  Stent Deployed: number analyzed (Participants) | 117
  Stent Deployed | 117

7. Secondary Outcome: Technical Success of Using the BRITE TIP RADIANZ™ Guiding Sheath
Description: Technical success associated with use of the BRITE TIP RADIANZ™ Guiding Sheath, defined as successful insertion of the device into the peripheral vasculature through the radial artery (allowing for introduction of interventional and/or diagnostic devices) and successful withdrawal of the device.
Time Frame: From the time of insertion through the time of withdrawal of the BRITE TIP RADIANZ™ Guiding Sheath through the radial access artery, assessed within the same day or 24 hours from the start time of the index procedure.
Population: Intent to Treat population of the main cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 129
Participants | 129

8. Secondary Outcome: Procedural Success of Using the SABERX RADIANZ™ PTA Balloon Catheter
Description: Procedural success associated with use of the SABERX RADIANZ™ PTA Balloon Catheter for pre-dilation and/or post-deployment stent dilatation (whenever applicable), defined as successful insertion of the device into the peripheral vasculature through the radial artery, successful inflation and deflation of the balloon, successful withdrawal of the device, and achievement of a final residual diameter stenosis of < 30% at the conclusion of the index procedure.
Time Frame: From the time of insertion to the time of withdrawal of the SABERX RADIANZ™ PTA Balloon Catheter through the radial access artery AND assessment of the final residual diameter stenosis, within the same day or 24 hours from the procedure start time
Population: There were 95 subjects with a complete set of available data to allow for endpoint analysis on the SABERX RADIANZ device.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 95
Participants | 79

9. Other Pre Specified Outcome: Fluoroscopy Time
Description: Fluoroscopy time is the length of time during which X-rays are produced during a fluoroscopy procedure.
Time Frame: From the start time to the end time of the period during which x-rays are produced, within the same day or 24 hours from the procedure start time
Population: Intent to Treat population of the main cohort
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interventional
Number analyzed (Participants) | 129
minutes | 9 (4)

10. Other Pre Specified Outcome: Time to Achieve Hemostasis
Description: Time to achieve hemostasis defined as the time elapsed from removal of the BRITE TIP RADIANZTM Guiding Sheath to the time that hemostasis was first observed.
Time Frame: From the time of removal of the BRITE TIP RADIANZ Guiding Sheath to when hemostasis was first observed, within the same day or 24 hours from the procedure start time
Population: Intent to Treat population of the main cohort
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interventional
Number analyzed (Participants) | 129
minutes | 47 (20)

11. Other Pre Specified Outcome: Time to Ambulation
Description: Time to ambulation, defined as the time from when vascular closure was achieved to when the subject could stand up and walk any distance
Time Frame: From the time of vascular closure to the time of ambulation, within the same day or 24 hours from the procedure start time, or study exit, whichever comes first
Population: Intent to Treat population of the main cohort. The Overall Number of Participants Analyzed is less than the total for the main cohort due to the unavailability of data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interventional
Number analyzed (Participants) | 40
minutes | 207 (153)

12. Other Pre Specified Outcome: Time to Hospital Discharge
Description: Time to hospital discharge
Time Frame: From the time of vascular closure to the time of hospital discharge (~ up to 1 week from date of index procedure) or study exit, whichever comes first
Population: Intent to Treat population of the main cohort. Outlier values noted for two subjects in the main cohort were removed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Interventional
Number analyzed (Participants) | 127
hours | 15.6 (9.5)

13. Other Pre Specified Outcome: Method to Achieve Closure of the Transradial Artery Access Site
Description: Method to achieve closure of the transradial artery access site
Time Frame: From the time of removing the BRITE TIP RADIANZ Guiding Sheath to the time of either removing the vascular closure device or ending manual compression, within the same day or 24 hours from the procedure start time
Population: Intent to Treat population of the main cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional
Number analyzed (Participants) | 129
Participants
  Manual Compression | 2
  Radial Compression Band | 127

14. Other Pre Specified Outcome: Quality of Life Assessed Via the SF-36 Questionnaires - General Health
Description: Mean scores are reported on a scale entitled "mean score" and range from 0 (minimum) to 100 (maximum); higher scores represent a better outcome.
Time Frame: Screening is up to 7 days prior to the index procedure date; discharge is between end of index procedure and 7 days post-discharge; the 30-day follow-up visit is between 23 and 37 days post-procedure, or until time of study exit (whichever comes first)
Population: Intent to Treat population of the main cohort
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional
Number analyzed (Participants) | 129
score on a scale
  Screening | 47.56 (17.67)
  Discharge | 52.44 (15.10)
  30 Day Follow-Up | 60.71 (16.43)

15. Other Pre Specified Outcome: Quality of Life Assessed Via the EuroQOL-5 Dimensions (EQ-5D) Questionnaire - Overall Health
Description: The EQ-5D questionnaire is an instrument designed to assess quality of life along five (5) dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. For each participant, a value-based scoring system is used to convert the combination of their responses to the five individual subscales into a single index value (or a code), which is then converted into a single score based on how people in the participant's country rate different combinations of problems.
  The EQ-5D score for Overall Health is reported as a mean and standard deviation at screening, discharge and 30 days in this module and ranges from 0 (minimum) to 100 (maximum) with higher scores representing better outcomes.
Time Frame: as for outcome 14
Population: Intent to Treat population of the main cohort
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional
Number analyzed (Participants) | 129
score on a scale
  Screening | 63.20 (16.24)
  Discharge | 70.66 (14.08)
  30 Day | 78.01 (13.95)

16. Other Pre Specified Outcome: Time to Hospital Discharge Eligibility
Description: Time to hospital discharge eligibility (when physician examines and if all is well, gives discharge orders)
Time Frame: From the time of vascular closure to the time of hospital discharge eligibility (~ up to 1 week from date of index procedure) or study exit, whichever comes first
Population: Intent to Treat population of the main cohort. The Overall Number of Participants Analyzed is less than the total number of participants in the main cohort due to the unavailability of data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Interventional
Number analyzed (Participants) | 39
hours | 14.3 (10.1)

17. Other Pre Specified Outcome: Procedural Time
Description: Procedural Time is defined as the time elapsed from when the sheath was introduced through the radial access artery to the time of vascular closure.
Time Frame: From the time of introduction of the sheath through the radial access artery to the time of vascular closure, within the same day or 24 hours from the procedure start time
Population: Intent to Treat population of the main cohort
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interventional
Number analyzed (Participants) | 129
minutes | 47 (20)

ADVERSE EVENTS:
Time Frame: Peri-procedural (within 30 days post-index procedure)
Groups:
- Main Cohort: The main cohort consisted of 129 of the 151 total enrolled subjects in the study.
- Roll-in Cohort: The roll-in cohort was a subgroup of 22 of the 151 total enrolled subjects. The roll-in cohort consisted of the first two (2) enrolled subjects at each study site (as applicable). Such subjects were pre-specified as "roll-in" subjects prior to their enrollment and met all criteria for enrollment, however, they were also followed up and evaluated up to 30 days post-procedure only for safety and not included in any primary endpoint analyses.
Arm/Group | Main Cohort | Roll-in Cohort
All-Cause Mortality (participants affected / at risk) | 0/129 | 1/22
Serious Adverse Events (participants affected / at risk) | 5/129 | 6/22
Other Adverse Events (participants affected / at risk) | 10/129 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort (N=129) | Roll-in Cohort (N=22)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Iliac artery perforation (Cardiac disorders) | 0 (0) | 1 (1)
Ulcer (General disorders) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort (N=129) | Roll-in Cohort (N=22)
Vascular access site haematoma (General disorders) | 10 (10) | 0 (0)

LIMITATIONS AND CAVEATS:
The cohort investigated excluded patients with various, pre-existing conditions and comorbidities, and so experienced clinicians should carefully consider in whom they prescribe intervention with the S.M.A.R.T. RADIANZ™ Vascular Stent System. Future studies could be undertaken to better ascertain the PAD patient cohorts that most likely stand to benefit from specifically from radial access and the S.M.A.R.T. RADIANZ™ Vascular Stent System compared to other contemporary treatment approaches.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication, provided that those comments do not jeopardize the scientific integrity of the publication.

DOCUMENTS (2):
  • Study Protocol (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT05399680/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT05399680/SAP_001.pdf